CLINICAL TRIAL: NCT07154147
Title: Cataract Oral vs IV Sedation Pilot RCT: A Non-inferiority Assessment of Perioperative Safety and Cognitive Recovery in Older Adults
Brief Title: Oral vs IV Sedation for Cataract Surgery in Older Adults
Acronym: CatNAPS-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-43837
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cataract Surgery; Sedation; Cognition Function; Perioperative Care; Older Adults
Keywords: oral sedation; intravenous sedation; alprazolam; midazolam; cataract surgery; older adults; cognitive recovery; postoperative recovery; patient satisfaction; non-inferiority trial; pilot study; randomized controlled trial; anesthesia
MeSH Terms: conditions — Patient Satisfaction | interventions — Alprazolam; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either oral sedation with IV placebo or IV sedation with oral placebo for cataract surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study. Participants, care providers (including surgeons and anesthesia teams), outcome assessors, and investigators will all be blinded to group assignment. Pharmacy staff managing randomization will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Sedation Group (Experimental): Participants in this group will receive oral sedation with alprazolam (0.5 mg) and IV placebo prior to cataract surgery. All participants will undergo standard cataract surgery with local anesthetic eye drops and continuous anesthesia monitoring. An IV line will be placed for monitoring, and anesthesia staff will be present during surgery, with the option to administer additional sedation if clinically indicated.
  Interventions: Drug: Alprazolam
- IV Sedation Group (Active Comparator): Participants in this group will receive IV sedation with midazolam (1 mg) and an oral placebo pill prior to cataract surgery. All participants will undergo standard cataract surgery with local anesthetic eye drops and continuous anesthesia monitoring. An IV line will be placed for monitoring, and anesthesia staff will be present during surgery, with the option to administer additional sedation if clinically indicated.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Alprazolam — Participants will take oral alprazolam 0.5 mg 15 to 90 minutes before surgery to promote relaxation and reduce anxiety. An IV placebo (normal saline) will be administered to maintain blinding.
  Other Names: Xanax
  Arms: Oral Sedation Group
Drug: Midazolam — Participants will receive IV midazolam 1 mg immediately before surgery to promote relaxation and reduce anxiety. An oral placebo pill will be used to maintain blinding.
  Other Names: Versed
  Arms: IV Sedation Group

SUMMARY:
The goal of this clinical trial is to find out if taking a pill (oral sedation) works just as well as getting medicine through a vein (IV sedation) to help older adults feel relaxed during cataract surgery. We are also studying how these two methods affect recovery, especially thinking and memory after surgery, and how satisfied people are with their care. Participants in this study will be randomly assigned to receive either oral sedation (+ IV placebo) or IV sedation (+ oral placebo) before their cataract surgery. They will complete short surveys about their thinking and recovery before and after surgery, and will be contacted by phone after surgery to check on their recovery. The results of this study will help doctors understand if a simple pill can be a safe and effective alternative to IV sedation for cataract surgery.

DETAILED DESCRIPTION:
This clinical trial is designed to compare two common ways of providing sedation during cataract surgery in older adults: oral sedation (a pill) and intravenous (IV) sedation (medicine given through a vein). Cataract surgery is a quick and safe procedure that helps people see better by removing the cloudy lens in their eye. While numbing eye drops are routinely used to prevent pain, many people also receive sedation to feel calm during surgery. In the United States, IV sedation is commonly used and requires close monitoring by an anesthesia team. In other countries, oral sedation is often used instead because it is simpler and less resource-intensive.

The goal of this study is to see if oral sedation can provide the same level of safety, comfort, and recovery as IV sedation. Researchers are especially interested in how each type of sedation affects a person's thinking, memory, and overall recovery in the days after surgery. The study also looks at how satisfied participants are with their care, whether they experience side effects, and whether surgeons feel the surgery goes smoothly with each type of sedation.

This is a small, pilot study that will enroll 20 adults aged 65 and older who are scheduled for cataract surgery. Participants will be randomly assigned by chance (like flipping a coin) to one of two groups: one group will receive a pill called alprazolam and a harmless IV placebo, while the other group will receive a placebo pill and standard IV sedation with a medication called midazolam. Everyone will still get numbing eye drops and be monitored by an anesthesia team during surgery for safety.

Participants will complete simple memory and recovery tests before and after surgery, and follow-up phone calls will check on how they are feeling up to seven days after surgery. By closely monitoring thinking ability, comfort, and safety, this study aims to provide important information about whether oral sedation could be a good option for people undergoing cataract surgery in the United States. The results will help guide future research and inform doctors about the best ways to care for older adults during eye surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 65 years old
2. Capable of providing informed consent and completing the study procedures in English
3. Able to provide consent for oneself
4. Able to follow directions
5. Able to climb one flight of stairs without stopping to rest
6. Have a new diagnosis of cataract disease
7. Plan on having cataract surgery on their eye within the next 6 months

Exclusion Criteria:

1. History of prior cataract surgery
2. Admission to the hospital within the past 30 days
3. Difficulty being sedated during other minor outpatient procedures or imaging studies
4. Allergy or resistance to local anesthetic agents
5. Cannot lay flat without having symptoms (i.e., difficulty breathing, severe back pain, etc.)
6. History of severe anxiety requiring routine use of benzodiazepines
7. Patient undergoing cataract surgery in combination with any other ophthalmologic procedure
8. Patient requiring general anesthesia during cataract surgery due to the underlying characteristics of the existing cataract and/or anticipated complexity of the planned procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with cognitive recovery based on the Postoperative Quality of Recovery Scale (PQRS) at multiple time points | before surgery, immediately after surgery, post-operative day 1, post-operative day 7
  Cognitive recovery will be measured using the cognitive domain of the PQRS, a validated questionnaire assessing recovery across several health domains. Recovery is defined by meeting pre-specified criteria for return to baseline cognitive function compared to pre-surgery testing

SECONDARY OUTCOMES:
Participant satisfaction with sedation experience using the Iowa Satisfaction with Anesthesia Scale (ISAS) | immediately after surgery, post-operative day 1, post-operative day 7
  Participants will complete the ISAS to rate satisfaction with their anesthesia experience, including feelings of relaxation, comfort, and recall of surgery
Surgeon Satisfaction with Intraoperative Conditions | Immediately after surgery
  Measured via post-surgery surgeon questionnaire assessing perceived ease of surgery, patient cooperation, and need for additional sedation
Feasibility of Recruitment | Throughout enrollment period
  Proportion of eligible participants who agree to participate in the trial
Participant Retention After Intervention | Up to 7 days post-surgery
  Proportion of enrolled participants who complete all postoperative follow-up assessments
Adherence to Sedation Intervention | Day of surgery
  Proportion of participants who receive their assigned intervention without protocol deviation (defined as receiving the intended oral or IV sedative)
Intervention Fidelity | Day of surgery
  Proportion of cases where study procedures were delivered as intended, including timing of medication administration and adherence to blinding protocol
Intraoperative Events | During surgery
  Incidence of intraoperative events, including: Participant complaints of pain or discomfort, anxiety or nervousness, requests for additional IV medication, undesirable patient movement, surgeon complaints about sedation adequacy, conversion to general anesthesia
Incidence of Postoperative Anesthesia-Related Complications | Up to 7 days after surgery
  Incidence of adverse events including delirium, nausea, vomiting, dizziness, falls, and unplanned healthcare utilization within 7 days post-surgery
Quality of Recovery Post-Surgery | Days 1 and 7 after surgery
  Measured by the Quality of Recovery domain of the PQRS (Postoperative Quality of Recovery Scale), including physical comfort, emotional well-being, and cognitive function compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Chen, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Wayne and Gladys Valley Center for Vision, Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a small single center pilot study so we do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Shah U, Wong D, Wong J. Patient satisfaction and positive patient outcomes in ambulatory anesthesia. Ambulatory Anesthesia. 2015;2:29-37 https://doi.org/10.2147/AA.S59820
- [Background] Kugler LJ, Kapeles MJ, Durrie DS. Safety of office-based lens surgery: U.S. multicenter study. J Cataract Refract Surg. 2023 Sep 1;49(9):907-911. doi: 10.1097/j.jcrs.0000000000001231. PMID 37276271
- [Background] Perumal D, Dudley RA, Gan S, Boscardin WJ, Gill A, Gelb AW, Lee SJ, Chen CL. Anesthesia Care for Cataract Surgery in Medicare Beneficiaries. JAMA Intern Med. 2022 Oct 3;182(11):1171-80. doi: 10.1001/jamainternmed.2022.4333. Online ahead of print. PMID 36190717
- [Background] Lee RM, Thompson JR, Eke T. Severe adverse events associated with local anaesthesia in cataract surgery: 1 year national survey of practice and complications in the UK. Br J Ophthalmol. 2016 Jun;100(6):772-6. doi: 10.1136/bjophthalmol-2015-307060. Epub 2015 Sep 24. PMID 26405103
- [Background] Ianchulev T, Litoff D, Ellinger D, Stiverson K, Packer M. Office-Based Cataract Surgery: Population Health Outcomes Study of More than 21 000 Cases in the United States. Ophthalmology. 2016 Apr;123(4):723-8. doi: 10.1016/j.ophtha.2015.12.020. Epub 2016 Jan 22. PMID 26804760
- [Background] Dexter F, Candiotti KA. Multicenter assessment of the Iowa Satisfaction with Anesthesia Scale, an instrument that measures patient satisfaction with monitored anesthesia care. Anesth Analg. 2011 Aug;113(2):364-8. doi: 10.1213/ANE.0b013e318217f804. Epub 2011 Apr 25. PMID 21519043
- [Background] Fung D, Cohen M, Stewart S, Davies A. Can the Iowa Satisfaction with Anesthesia Scale be used to measure patient satisfaction with cataract care under topical local anesthesia and monitored sedation at a community hospital? Anesth Analg. 2005 Jun;100(6):1637-1643. doi: 10.1213/01.ANE.0000154203.00434.23. PMID 15920188
- [Background] Katz J, Feldman MA, Bass EB, Lubomski LH, Tielsch JM, Petty BG, Fleisher LA, Schein OD; Study of Medical Testing for Cataract Surgery Study Team. Adverse intraoperative medical events and their association with anesthesia management strategies in cataract surgery. Ophthalmology. 2001 Oct;108(10):1721-6. doi: 10.1016/s0161-6420(01)00704-7. PMID 11581040
- [Background] Norregaard JC, Schein OD, Bellan L, Black C, Alonso J, Bernth-Petersen P, Dunn E, Andersen TF, Espallargues M, Anderson GF. International variation in anesthesia care during cataract surgery: results from the International Cataract Surgery Outcomes Study. Arch Ophthalmol. 1997 Oct;115(10):1304-8. doi: 10.1001/archopht.1997.01100160474016. PMID 9338678
- [Background] Peeler CE, Villani CM, Fiorello MG, Lee HJ, Subramanian ML; Oral versus Intravenous Sedation Study Group. Patient Satisfaction with Oral versus Intravenous Sedation for Cataract Surgery: A Randomized Clinical Trial. Ophthalmology. 2019 Sep;126(9):1212-1218. doi: 10.1016/j.ophtha.2019.04.022. Epub 2019 Apr 16. PMID 31002834
- [Background] Chen CL, Lin GA, Bardach NS, Clay TH, Boscardin WJ, Gelb AW, Maze M, Gropper MA, Dudley RA. Preoperative medical testing in Medicare patients undergoing cataract surgery. N Engl J Med. 2015 Apr 16;372(16):1530-8. doi: 10.1056/NEJMsa1410846. PMID 25875258